CLINICAL TRIAL: NCT07405528
Title: Camouflaged WeChat Mini-program-based Intervention for Women Victims of Intimate Partner Violence: Protocol for a Pilot Mixed Methods Study
Brief Title: Camouflaged WeChat-based Intervention for Abused Women
Acronym: IPV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22232811; 22232811 (Other Grant/Funding Number: Health and Medical Research Fund)
Record Dates: First submitted 2025-12-29; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Domestic Violence; Mental Health Wellness 1
Keywords: Domestic Violence; Intimate partner violence; mHealth intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WOMEN Health group (Experimental): The WOMEN Health programme
  Interventions: Behavioral: WOMEN Health programme
- Wait-list control group (Active Comparator): Healthy lifestyle intervention
  Interventions: Behavioral: Wait-list control group

INTERVENTIONS:
Behavioral: WOMEN Health programme — (i) Empowerment (IPV information, ie, 30-min one-to-one interview, WeChat mini-program); (ii) Telephone social support (ie, weekly calls); (ⅲ) Healthy lifestyle intervention (ie, healthy lifestyle information and discussion)
  Arms: WOMEN Health group
Behavioral: Wait-list control group — (i) Healthy lifestyle intervention (ie, discussion and weekly calls for body weight)
  Arms: Wait-list control group

SUMMARY:
Intimate partner violence (IPV) is a major public health issue and human rights threat worldwide, especially for Chinese immigrant women victims in Hong Kong. Interventions that address negative physical and emotional outcomes from IPV could therefore play a crucial role in enhancing empowerment, social support, and healthy lifestyle among these women. The overall objective of this pilot mixed methods study is to determine the feasibility and acceptability of a camouflaged WeChat mini-program-based WOMEN Health intervention for women victims of IPV. This study will evaluate the feasibility and acceptability of a camouflaged WeChat mini-program-based WOMEN Health intervention for women victims of IPV.

DETAILED DESCRIPTION:
Intimate partner violence (IPV) is a major public health issue and human rights threat worldwide, especially for Chinese immigrant women victims in Hong Kong. Interventions that address negative physical and emotional outcomes from IPV could therefore play a crucial role in enhancing empowerment, social support, and healthy lifestyle among these women. Previous studies in Hong Kong and the United States provided evidence on IPV interventions among Chinese abused women; however, there is a scarcity of evidence on the use of mHealth for abused women while fully considering their safety studies on mobile technology for Chinese immigrant women victims are limited, and there lacks safe, low-cost, and evidence-based mHealth interventions for empowering and supporting women victims who immigrate to Hong Kong and face more vulnerabilities and needs. This study will evaluate the feasibility and acceptability of a camouflaged WeChat mini-program-based WOMEN Health intervention for women victims of IPV.

This pilot mixed methods study will adopt the randomized, wait-list controlled trial with two groups (1:1 ratio), followed by in-depth interviews with participants in the WOMEN Health programme group at post-intervention. It will evaluate feasibility and acceptability as the primary outcomes and compare scores changes after 12 weeks interventions between Chinese immigrant women who are screened positive for IPV randomly assigned to receiving genuine IPV intervention and disguised healthy lifestyle intervention, and Chinese immigrant women who are screened positive for IPV in a control procedure. The wait-list control group will also receive the WOMEN Health programme after the intervention group completed the programme.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese-speaking (Mandarin or Cantonese)
2. women aged 18 to 45 years
3. originally from mainland China and have moved to Hong Kong for at least one year
4. screened positive for IPV during heterosexual relationships in the past year
5. have a smartphone with WeChat installed
6. with no plans to move outside Hong Kong in the next one year

Exclusion Criteria:

1. unwilling to provide informed consent
2. severe chronic diseases (e.g., cancer, heart failure, kidney failure, chronic obstructive pulmonary disease, and HIV/AIDS)
3. currently experience severe IPV (identified using the revised 11-item Danger Assessment)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 86 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of the WOMEN Health programme | Week 12
  Feasibility and acceptability will be assessed using a 12-item self-developed questionnaire. Items are rated on a 5-point Likert scale (1-5), with higher scores indicating greater acceptability, satisfaction, and usefulness.

SECONDARY OUTCOMES:
Changes in depressive symptoms | Baseline and Week 12
  Depressive symptoms will be assessed using the Chinese version of the Beck Depression Inventory-II (BDI-II), a 21-item self-report questionnaire measuring depressive symptoms experienced over the past two weeks. Total scores range from 0 to 63, with higher scores indicating more severe depressive symptoms.
Changes in quality of life | Baseline and Week 12
  Quality of life will be assessed using the Chinese version of the 12-Item Short Form Health Survey, version 2 (SF-12v2), which measures physical and mental health status. Physical Component Summary (PCS) and Mental Component Summary (MCS) scores range from 0 to 100, with higher scores indicating better quality of life.
Changes in intimate partner violence (IPV) | Baseline and Week 12
  Intimate partner violence will be assessed using the Chinese version of the Revised Conflict Tactics Scales (CTS2), which measures the frequency and severity of psychological aggression, physical assault, sexual coercion, and injury within intimate relationships. Higher scores indicate greater exposure to intimate partner violence.
Changes in Body Mass Index (BMI) | Baseline and up to 12 weeks
  Body weight will be self-measured by participants at home in the morning under fasting conditions, wearing light clothing and without shoes. Height will be measured at baseline using a wall-mounted stadiometer. BMI will be calculated as body weight in kilograms divided by height in meters squared (kg/m²) and categorized according to the World Health Organization (WHO) recommendations for Asian populations.
Changes in healthy behaviors | Baseline and Week 12
  Healthy lifestyle behaviors, including physical activity and dietary behaviors, will be documented by self-report data

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Draughon Moret J, Todd A, Rose L, Pollitt E, Anderson J. Mobile Phone Apps for Intimate Partner and Sexual Violence Prevention and Response: Systematic Search on App Stores. JMIR Form Res. Feb 8 2022;6(2):e28959. doi:10.2196/28959
- [Result] Glass NE, Clough A, Messing JT, et al. Longitudinal Impact of the myPlan App on Health and Safety Among College Women Experiencing Partner Violence. J Interpers Violence. Jul 2022;37(13-14):Np11436-np11459. doi:10.1177/0886260521991880
- [Result] Lin Z, Cheng L, Han X, et al. The Effect of Internet-Based Cognitive Behavioral Therapy on Major Depressive Disorder: Randomized Controlled Trial. J Med Internet Res. Sep 22 2023;25:e42786. doi:10.2196/42786
- [Result] Chen D, Zhang H, Wu J, et al. Effects of an Individualized mHealth-Based Intervention on Health Behavior Change and Cardiovascular Risk Among People With Metabolic Syndrome Based on the Behavior Change Wheel: Quasi-Experimental Study. J Med Internet Res. Nov 29 2023;25:e49257. doi:10.2196/49257
- [Result] Sumra M, Asghar S, Khan KS, Fernández-Luna JM, Huete JF, Bueno-Cavanillas A. Smartphone Apps for Domestic Violence Prevention: A Systematic Review. Int J Environ Res Public Health. Mar 23 2023;20(7)doi:10.3390/ijerph20075246
- [Result] Tong A, Sainsbury P, Craig J. Consolidated criteria for reporting qualitative research (COREQ): a 32-item checklist for interviews and focus groups. Int J Qual Health Care. 2007 Dec;19(6):349-57. doi: 10.1093/intqhc/mzm042. Epub 2007 Sep 14. PMID 17872937
- [Result] Li Y, Rhee H, Bullock LFC, McCaw B, Bloom T. Self-Compassion, Health, and Empowerment: A Pilot Randomized Controlled Trial for Chinese Immigrant Women Experiencing Intimate Partner Violence. J Interpers Violence. 2024 Apr;39(7-8):1571-1595. doi: 10.1177/08862605231207624. Epub 2023 Oct 30. PMID 37902465
- [Result] Chan KL. Correlates of wife assault in Hong Kong Chinese families. Violence Vict. Apr 2004;19(2):189-201. doi:10.1891/vivi.19.2.189.64104
- [Result] Barbara MB, S. SM, H. PW. Validating the Beck Depression Inventory-II for Hong Kong Community Adolescents. International Journal of Testing. 2004;4(3):199-216. doi:10.1207/s15327574ijt0403_1
- [Result] Tiwari A, Leung WC, Leung TW, Humphreys J, Parker B, Ho PC. A randomised controlled trial of empowerment training for Chinese abused pregnant women in Hong Kong. Bjog. Sep 2005;112(9):1249-56. doi:10.1111/j.1471-0528.2005.00709.x
- [Result] Tiwari A, Fong DYT, Yuen FKH, Fung HYK, Pang POY, Wong JYH. Purpose-built intervention for mental health of Mainland Chinese immigrant women survivors of intimate partner violence: a randomised controlled trial (abridged secondary publication). Hong Kong Med J. 2020 Dec;26 Suppl 8(6):7-9. No abstract available. PMID 33504670
- [Result] Broadhurst R, Bouhours B, Bacon-Shone J. Hong Kong the international violence against women survey: final report of the 2006 Hong Kong IVAWS. 2012. doi.org/10.2139/ssrn.2076994.

DOCUMENTS (1):
  • Informed Consent Form (2024-12-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT07405528/ICF_000.pdf